CLINICAL TRIAL: NCT06664866
Title: Artificial Intelligence Guided Echocardiographic Screening of Rare Diseases (EchoNet-Screening)
Brief Title: AI Echocardiographic Screening of Cardiac Amyloidosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Palo Alto Veteran Affairs Hospital (Unknown); Providence Heart & Vascular Institute (Other); Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Lily Stern, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Study1720
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Suspicious by EchoNet-LVH Algorithm (Experimental): Each potential participant identified by automated AI-enhanced echocardiogram review will be chart reviewed by each site's CA experts for appropriateness of enrollment and clinican suspicion for CA. Based on the judgement of CA experts, potential participants that meet eligibility criteria will be called to be consented, followed in the study, and referred to see the CA expert.
  Interventions: Diagnostic Test: EchoNet-LVH Assessment

INTERVENTIONS:
Diagnostic Test: EchoNet-LVH Assessment — The AI algorithm is previously described (Duffy et al. JAMA Cardiology 2022) and will remain unchanged throughout the course of the study. A pre-determined threshold based on prior experiments and analysis has been decided prior to the study. From each site, approximately 100,000 echocardiogram studies will be reviewed by EchoNet-LVH for approximately 500 patients to be flagged.

SUMMARY:
Recent advances in machine learning and image processing techniques have shown that machine learning models can identify features unrecognized by human experts and accurately assess common measurements made in clinical practice. Echocardiography is the most common form of cardiac imaging and is routinely and frequently used for diagnosis. However, there is often subjectivity and heterogeneity in interpretation. Artificial intelligence (AI)'s ability for precision measurement and detection is important in both disease screening as well as diagnosis of cardiovascular disease.

Cardiac amyloidosis (CA) is a rare, underdiagnosed disease with targeted therapies that reduce morbidity and increase life expectancy. However, CA is frequently overlooked and confused with heart failure with preserved ejection fraction. Some estimates suggest that CA can be as prevalence as 1% in a general population, with even higher prevalence in patients with left ventricular hypertrophy, heart failure, and other cardiac symptoms that might prompt echocardiography.

AI guided disease screening workflows have been proposed for rare diseases such as cardiac amyloidosis and other diseases with relatively low prevalence but significant human impact with targeted therapies when detected early. This is an area particularly suitable for AI as there are multiple mimics where diseases like hypertrophic cardiomyopathy, cardiac amyloidosis, aortic stenosis, and other phenotypes might visually be similar but can be distinguished by AI algorithms. The investigators have developed an algorithm, termed EchoNet-LVH, to identify cardiac hypertrophy and identify patients who would benefit from additional screening for cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving an echocardiogram that is determined to be suspicious by EchoNet-LVH

Exclusion Criteria:

* Patients that decline consent
* Patients receiving an echocardiogram that is determined to be not suspicious by EchoNet-LVH

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value | 1 year
  1. Among patients that screening positive and consented to the trial, the proportion of patients that subsequently are confirmed to have CA upon clinical follow-up.
  2. Statistical Analysis: Fisher's exact (two-sided) for superiority Comparison with PPV of standard clinical suspicion (PPV of all comers that receive Tc-99m PYP/HDP imaging scan or other clinical diagnosis).

SECONDARY OUTCOMES:
Time to Diagnosis from Echocardiogram Study to Clinical Diagnosis | 1 year
  Statistical Analysis: Cox proportional hazards test with comparison with of Study population vs. comparison with Patients with echocardiogram study showing at least moderate left ventricular hypertrophy by human interpretation.
Number of Patients that Receive Treatment for CA | 1 year
Number of Cardiac Amyloidosis Diagnoses | 1 year
Number of Participants with All Cause Death | 1 year
Number of Participants with All Cause Hospitalization | 1 year
Number of Participants with Heart Failure Hospitalization | 1 year
  defined as needing IV diuretics or BNP higher than baseline or ICD9/10 code

CONTACTS AND LOCATIONS:
Overall Officials: Lily Stern, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (4):
- United States (4):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Palo Alto Veteran Affairs Hospital, Palo Alto, California
  - Northwestern Medicine, Chicago, Illinois
  - Providence Heart and Vascular Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No